CLINICAL TRIAL: NCT00986401
Title: Safety and Tolerability of Trospium Chloride Metformin Hydrochloride in Healthy Subjects
Brief Title: Safety and Tolerability of Trospium Chloride and Metformin Hydrochloride in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MA-SXR-09-002
Record Dates: First submitted 2009-09-16; First posted 2009-09-30 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Adults
MeSH Terms: interventions — trospium chloride; Metformin

ARMS (2):
- Glucophage® then Sanctura XR® (AB) (Experimental): Treatment Period 1: Glucophage® (500 mg, BID) for 3.5 days. Washout: There will be a washout period of 3 days between each treatment period. Treatment Period 2: Sanctura XR® (60 mg, QD) for 10 days followed by Sanctura XR® (60 mg, QD) for 4 days + Glucophage® (500 mg, BID) for 3.5 days.
  Interventions: Drug: Metformin hydrochloride (Glucophage®)
- Sanctura XR® then Glucophage® (BA) (Experimental): Treatment Period 1: Sanctura XR® (60 mg, QD) for 10 days followed by Sanctura XR® (60 mg, QD for 4 days) + Glucophage® (500 mg, BID) for 3.5 days. Washout: There will be a washout period of 3 days between each treatment period. Treatment Period 2: Glucophage® (500 mg, BID) for 3.5 days.
  Interventions: Drug: Trospium Chloride (Sanctura XR®)

INTERVENTIONS:
Drug: Trospium Chloride (Sanctura XR®) — extended release, 60 mg, oral daily
  Other Names: Sanctura XR® 60 mg
  Arms: Sanctura XR® then Glucophage® (BA)
Drug: Metformin hydrochloride (Glucophage®) — immediate release, 500mg
  Other Names: Glucophage®
  Arms: Glucophage® then Sanctura XR® (AB)

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of trospium chloride (Sanctura XR™) and metformin hydrochloride (Glucophage) when co-administered.

ELIGIBILITY:
Inclusion Criteria:

* Weight within +/-30% of ideal body weight for height and frame size
* Non-smoker (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 1 months prior to the screening visit).
* Willing to abstain from caffeine-containing food and beverages for 24-hours prior to dosing, alcohol-containing food and beverage for 48 hours prior to dosing, and Seville oranges (eg orange marmalade), grapefruit, or grapefruit juice for 7 days prior to the dosing and abstain from all throughout the study.
* Willing to abstain from taking medications (with the exception of hormonal contraceptives) and nonprescription medication including vitamins, food supplements, and herbal preparations for 7 days prior to Day-1 of the first treatment period and throughout the study.

Exclusion Criteria:

* Uncontrolled systemic disease
* Known allergy or sensitivity to the study medication(s) (Trospium, Metformin)or its components
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* History of myasthenia gravis or closed-angle glaucoma.
* Considering or scheduled to undergo any surgical procedure during the study.
* History of alcohol or substance abuse within 1 year prior to Day-1 of the first treatment period.
* History of serious mental or physical illness.
* Donated in excess of 500 mL of blood in the 30 days prior to the screening visit.
* Required treatment with any medications, either prescription or nonprescription (including vitamins, antacids, acid-reducers, food supplements, and herbal preparations, excluding hormonal contraceptives), within 7 days prior to Day-1 of the first treatment period during the study.
* Had an acute illness within 5 days prior to Day-1 of the treatment period.
* Had a history of hepatitis B or C, a positive test for hepatitis B surface antigen, hepatitis C antibody, a history of human immunodeficiency virus (HIV) infection or demonstration of HIV antibodies.
* Planned radiologic study requiring intravenous contrast administration of iodinated contrast material during the study period Serum Creatinine greater than 1.4 mg/dL.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Glucophage® Then Sanctura XR® (AB) | Sanctura XR® Then Glucophage® (BA)
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Period: Period 2
Arm/Group | Glucophage® Then Sanctura XR® (AB) | Sanctura XR® Then Glucophage® (BA)
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucophage® Then Sanctura XR® (AB) | Sanctura XR® Then Glucophage® (BA) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age Continuous [Median (Full Range); unit: years] | 31.0 [18 to 44] | 30.2 [18 to 44] | 31.0 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Level (Cmax) of Metformin Hydrochloride (Glucophage®) Following Oral Administration of Glucophage®
Description: Maximum Plasma Level (Cmax) of Metformin Hydrochloride (Glucophage®) following oral administration of Glucophage® alone and in combination with SanturaXR®. Plasma is the fluid portion of the blood.
Time Frame: 34 Days
Population: Intent-to-treat, which includes all patients who started the study (randomized). One patient was not included in the analysis due to early discontinuation.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Groups:
- Glucophage®: Glucophage®
- Glucophage® + Sanctura XR®: Glucophage® + Sanctura XR®
Arm/Group | Glucophage® | Glucophage® + Sanctura XR®
Number analyzed (Participants) | 43 | 43
Nanograms per milliliter (ng/mL) | 739 (263) | 753 (252)

2. Secondary Outcome: Maximum Plasma Level (Cmax) of Trospium Chloride (Sanctura XR®) Following Oral Administration of Sanctura XR®
Description: Maximum Plasma Level (Cmax) of Trospium Chloride (Sanctura XR®) Following Oral Administration of Sanctura XR® alone and in combination with Glucophage®. Plasma is the fluid portion of the blood in which the cells are suspended.
Time Frame: 34 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Groups:
- Sanctura XR®: Sanctura XR®
- Sanctura XR® + Glucophage®: Sanctura XR® + Glucophage®
Arm/Group | Sanctura XR® | Sanctura XR® + Glucophage®
Number analyzed (Participants) | 44 | 43
Nanograms per milliliter (ng/mL) | 1.87 (1.44) | 1.17 (0.71)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated.
Groups:
- Sanctura XR® in Combination With Glucophage®: Sanctura XR® in combination with Glucophage®
Arm/Group | Glucophage® | Sanctura XR® | Sanctura XR® in Combination With Glucophage®
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 10/43 | 3/44 | 13/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glucophage® (N=43) | Sanctura XR® (N=44) | Sanctura XR® in Combination With Glucophage® (N=44)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 4 | 3 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No